CLINICAL TRIAL: NCT06029504
Title: Optical Guided Sentinel Node Biopsy for Staging of Vulvar Cancer
Brief Title: Optical Guided Sentinel Node Biopsy for Staging of Vulvar Cancer (I)
Acronym: SENTIVUC
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Ligita Paskeviciute Froding, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: H-18020235
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-09

CONDITIONS: Vulvar Cancer; Sentinel Lymph Node
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate whether Sentinel Node biopsy can be performed without the use of lymphoscintigraphy and with ICG as a mono-tracer in women with vulvar cancer, unifocal tumor < 4 cm (clinical stage IB and II). Further, to investigate the accuracy of combined PET-CT and ultrasound (US) of the groins with US-guided biopsy of suspicious lymph nodes for the identification of macro-metastases in women with vulvar cancer, unifocal tumor < 4 cm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary vulva cancer, FIGO stage IB (tumor < 4 cm)
* Patients with unifocal recurrence in the vulva (tumor < 4 cm) located on the side where the patient is surgically naïve in the groin

Exclusion Criteria:

* Prior irradiation of the vulva or groins
* Prior SNB or inguinal lymphadenectomy in the relevant groin
* Known allergy to ICG or iodine (ICG contains 5% sodium iodine)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary or recurrent vulva cancer
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sentinel Node detection rate | Three years
  SN detection rate with ICG and 99mTc-Nanocoll alone perioperatively, where lymphoscintigraphy is blinded, in patients with vulvar cancer (tumor < 4 cm) without clinical suspicion of metastases to the inguinal lymph nodes.

SECONDARY OUTCOMES:
Sensitivity, specificity, PPV and NPV | Three years
  Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of FDG PET-CT and US combined with US-guided biopsy of suspicious lymph nodes for the identification of macro-metastases in the groins

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital, Copenhagen, Denmark